CLINICAL TRIAL: NCT02002663
Title: Efficacy of the Intralesional Infusion of Local Anesthetic and Steroids After Major Abdominal Surgery: a Randomized Double Blind Phase III Trial
Brief Title: Continuous Local Anesthetic and Steroid Infusion in Abdominal Surgery
Acronym: GR-CWI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Massimo Allegri, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PT-SM-13- YR FIRST STEP CWI-PP
Record Dates: First submitted 2013-10-24; First posted 2013-12-06 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain | interventions — Methylprednisolone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ropivacaine + methylprednisolone (Experimental): Continuous infusion of Ropivacaine 0.2% and methylprednisolone 1mg/kg 10ml/h through intralesional catheter for 24 hours
  Interventions: Drug: ropivacaine 0.2%; Drug: Methylprednisolone 1mg/kg
- saline (Placebo Comparator): Continuous infusion of saline through intralesional catheter for 24 hs
  Interventions: Drug: saline 0.9%

INTERVENTIONS:
Drug: ropivacaine 0.2% — PCA morphine 0.5 mg/ml bolus 1 mg LO 5 min max 20 mg in 4 hs
  Other Names: morphine PCA
  Arms: ropivacaine + methylprednisolone
Drug: Methylprednisolone 1mg/kg
  Arms: ropivacaine + methylprednisolone
Drug: saline 0.9%
  Arms: saline

SUMMARY:
The aim of the study is the identification, comparing continuous infusion of local anesthetics and steroids intralesionally with the current gold standard therapy (PCA), of the effective dose of local anesthetics and steroids within 7 days following abdominal surgery in order to halve the consumption of opioids and give the best pain control with a lower incidence of side effects and persistent chronic pain (at 1 and 3 months) We also plan to measure the peripheral inflammation and oxidative stress by analyzing the pro-inflammatory cytokines and anti-inflammatory properties.

Another objective is to investigate the combined effect of polymorphisms of genes related to pain sensitivity, and the correlation with the development of the inflammatory response and the incidence of chronic post-surgical pain (CPSP), which will be considered to validate the genotype-phenotype correlations.

The intralesional catheter will be placed within the operating field by the surgeon at the end of the procedure.

* first postoperative 24 hours: ropivacaine 0.2%-methylprednisolone 1 mg/kg/die infusion (10ml/h) in the wound. Rescue dose with morphine via intravenous PCA (0.5 mg/ml, bolus 1 mg, lock-out 5 min, max 20 mg in 4 hours)
* from 24 hs to 48 hs: ropivacaine 0.2%-methylprednisolone 1 mg/kg/die infusion (10ml/h) or saline 0.9% 10 ml/h in the wound. Rescue dose with morphine via intravenous PCA (0.5 mg/ml, bolus 1 mg, lock-out 5 min, max 20 mg in 4 hours) . from 48 hs to 7th day: ropivacaine 0.2% or saline 0.9% via patient controlled intralesional analgesia (PCIA) (2 mg/ml, bolus 20 mg, lock-out 60 min, max 80 mg in 4 hours). Rescue dose Tramadol 100 mg.

The first assessment will be by the anesthetist pre-operatively, to verify the patient eligibility.

All patients will be evaluated at the end of surgery (T0) and after 3-6-12-24-36-48 hours after surgery. Further evaluations are scheduled every 24 hours until the seventh postoperative day. At each assessment will be recorded: Numeric Rating Scale (NRS) at rest, NRS at movement (NRSm) - defined as pain at deep inspiration and cough - ; blood pressure, heart rate, respiratory rate, nausea (PONV scale), need of rescue analgesics and presence of any complications.

On the 7th postoperative day, the patient will be reassessed by both pain clinicians and surgeon; the surgeon will remove the catheter.

At 1 month and 3 months after surgery, the patient will be evaluated through phone interview to investigate pain persistence.

Inflammatory response analysis will be performed on the first 15 patients in each group (for a total of 30 patients). Before awakening of the patient the surgeon will insert a microdialysis catheter in the fat adjacent to the surgical wound with sterile technique. The microdialysed liquid will be collected in dedicated tubes directly in the infusion pump. The sample of the first hour will be discarded to avoid that microtrauma of catheter positioning influences the study. Sampling will be performed every 6 hours the first day, and every 12 hours in the second and third day. Serum samples will be collected to compare systemic with regional samples. All samples will be stored at -80 ° C until sampling. Concentrations quantification of different cytokines will be analyzed by ELISA Parma Unit will analyze VNTR (variable number of tandem repeats) polymorphism of the ADRB2 gene, directly related to the risk of chronic persistent postoperative pain development; Pavia Unit will take care of genotyping of polymorphic sites in the following genes: OPRM1 (mu-opioid receptor 1), COMT (catecholamine O-methyl transferase), UGT2B7 (UDP-glucuronyl transferase), IL1Ra (interleukin 1receptor alpha). From the blood samples will be extracted DNA and RNA using standard procedures. RNA will be retained for possible future studies on the expression of genes of interest. The DNA will be used instead for the study of genetic polymorphisms.

In this study the formation of free radicals, particularly superoxide will be assessed together with lipid peroxidation in both serum and urine, The 8- deoxyguanosine and Poly-ADP-ribose polymerase (PARP), the presence of nitrotyrosine.

Blood samples and urine tests will be carried out before the start of surgery , before the bolus of morphine and local anesthetic , at 24 h after the end of the intervention and 48 h after end of the intervention

ELIGIBILITY:
Inclusion Criteria:

* Male and females 18-85 years old scheduled to use PCA with morphine for postoperative pain control
* HIV-negative
* Classification American Society of Anesthesiologists (ASA) I: without systemic disease
* Classification ASA II or III (moderate systemic disease or severe systemic disease that limits activity without disability)
* Scheduled for major abdominal and urologic surgery (no emergency surgery)

Exclusion Criteria:

* regular use of opioid analgesics;
* History of abuse of drugs and / or alcohol;
* Postoperative hospitalization in intensive care with sedation and / or mechanical ventilation;
* severe renal impairment (creatinine> 2 g / dl, creatinine clearance <30 ml / h) and / or hepatic impairment (cholinesterase <2000 IU);
* Cardiac disorders (arrhythmias, heart failure);
* Neurological disorders (epilepsy);
* Cognitive disorders, mental retardation, psychiatric disorders;
* Changes in the normal coagulation or coagulopathy (INR> 2, PTT> 44 sec);
* Platelet count less than 100.000/mm3;
* BMI> 30;
* Allergy to study drugs.
* diabetes type I/II

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-08; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
total morphine consumption | 7 days after surgery

SECONDARY OUTCOMES:
pain values | 7 days
  number of patients presenting NRS values lower than 4 both at rest and at movement
number of patients presenting methylprednisolone side effects | up to 7 days
  wound healing retardation or other side effects which could be related to steroid wound infusion
number of patients presenting morphine or ropivacaine side effects | up to 7 days
  incidence of PONV, pruritus and sedation; side effects related to local anesthetic's systemic absorption
persistent pain at 1 and 3 months | 3 months
  number of participants developing pain at 1 and 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - •2nd Service of Anesthesia, Intensive Care and Pain Therapy, University Hospital of Parma, Parma
  - Department of Anesthesia and ICU, General Surgery and Urology, S Matteo Hospital, Pavia

REFERENCES:
- [Derived] Bugada D, De Gregori M, Compagnone C, Muscoli C, Raimondi F, Bettinelli S, Avanzini MA, Cobianchi L, Peloso A, Baciarello M, Dagostino C, Giancotti LA, Ilari S, Lauro F, Grimaldi S, Tasciotti E, Fini M, Saccani Jotti GM, Meschi T, Fanelli G, Allegri M. Continuous wound infusion of local anesthetic and steroid after major abdominal surgery: study protocol for a randomized controlled trial. Trials. 2015 Aug 14;16:357. doi: 10.1186/s13063-015-0874-z. PMID 26272452